CLINICAL TRIAL: NCT07098728
Title: Intravenous Levetiracetam Versus Intravenous Phenobarbital in Children With Prolonged Seizures Unresponsive to Benzodiazepines
Brief Title: Levetiracetam Versus Phenobarbital in Benzodiazepines Unresponsive Paediatric Prolonged Seizures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ministry of Health and Sports, Myanmar (Other Government)
Responsible Party: Principal Investigator, Aung Kyaw Min, Consultant Paediatrician, Ministry of Health and Sports, Myanmar
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 55/UM1,REC.2024; Research and Ethics Committee (Other: University of Medicine 1, Yangon)
Record Dates: First submitted 2025-07-21; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2024-12

CONDITIONS: Seizure
Keywords: Status Epilepticus
MeSH Terms: conditions — Seizures; Status Epilepticus | interventions — Phenobarbital

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Injection Levetiracetam Group (Active Comparator): Injection Levetiracetam
  Interventions: Drug: Levetiracetam IV
- Injection Phenobarbital Group (Active Comparator): Injection Phenobarbital
  Interventions: Drug: Phenobarbital

INTERVENTIONS:
Drug: Levetiracetam IV — Leveget injection 500mg/5ml
  Arms: Injection Levetiracetam Group
Drug: Phenobarbital — Phenobarbital injection 200mg/ml (BPI Insein)
  Arms: Injection Phenobarbital Group

SUMMARY:
Convulsive prolonged seizures in children are the most common life-threatening neurological emergencies. The aim of active management of seizure control is to prevent irreversible neuronal damage as early as possible. Although there is evidence of the use of benzodiazepines as the initial management for prolonged seizures, up to a third of patients do not respond to benzodiazepines. Many trials study the rate of seizures control among various second-line antiseizure medications (ASMs) in benzodiazepines unresponsive convulsive prolonged seizures. However, there is still few recommendations for paediatric population which drug is the most effective to control seizures rapidly and there is also a limited data on which drug has less adverse effects and is well tolerated. Currently, injection phenobarbital or levetiracetam is used as second-line antiseizure medication based on expert opinion in many centres globally including Yangon Children's Hospital. From this study, it is expected to identify the safer and more effective second-line treatment for prolonged seizures in children and be helpful in considering the alternative choice of appropriate medications in the management of prolonged seizures to include in the local guideline. A hospital-based randomized comparative study will be conducted at Yangon Children's Hospital. All children with benzodiazepines unresponsive prolonged seizures will be eligible for this study with the minimum sample size of 180 (90:90). Consecutive sample collection by block randomization will be done throughout the study period. The informed consent will be taken after explanation of nature, purposes, procedure, durations, benefits and risks. This study will be started with the approval of Academic Board of Study and Research and Ethics Committee, University of Medicine 1, Yangon. By this study, clinical response of intravenous levetiracetam versus intravenous phenobarbital in children with benzodiazepines unresponsive prolonged seizures will be evaluated. Aim of this study is to study the clinical response of intravenous levetiracetam versus intravenous phenobarbital in children with prolonged seizures unresponsive to benzodiazepines. Findings will support the choice of the safer and more effective second-line treatment for prolonged seizures in Myanmar children.

After case selection according to inclusion criteria and getting informed consent, computerized block randomization will be done. Total 9 blocks will be generated with group A and group B. Each child will be assigned as group A or group B according to randomization. All patients will be received supportive care according to treatment guideline of the ward. Group A patients will be treated with intravenous levetiracetam 40 mg/kg (maximum of 3000 mg) over 15 minutes. Group B patients will be treated with intravenous phenobarbital 20 mg/kg (maximum of 1000 mg) over 20 minutes. Injection levetiracetam will be diluted with 5% dextrose water to a concentration of 50 mg/ml. Injection phenobarbital will be diluted to become 20 ml with 5% dextrose water. All participants will also be monitored for oxygen saturation, respiratory rate and pattern, pulse rate, pulse volume, and blood pressure to detect treatment-related adverse effects. Monitoring will be conducted before, during, and 5 minutes after the assigned drug infusion, then hourly for 4 hours, every 2 hours for the following 4 hours, and every 4 hours thereafter.

The primary outcome of the study will be the clinical cessation of the seizure at five minutes after the completion of the infusion of intravenous levetiracetam or phenobarbital. The secondary outcome of the study will be the recurrence of seizure within 12 hours after the commencement of the study medications, need of other medications for active seizure control within 12 hours after the commencement of the study medications, need for rapid sequence induction (RSI) with thiopentone for on-going seizure management after administration of study medications. These secondary outcomes will be assessed in treatment-responsive groups. Treatment related adverse effects will also be assessed within five minutes of drug infusion in both treatment groups and within 12 hours in treatment-responsive groups. Data analysis will be done to compare the clinical response.

If the patient's seizure has stopped five minutes after completing the infusion of the assigned medication, a maintenance dose of either levetiracetam or phenobarbital, whichever was previously used, will be administered intravenously. If the patient is still experiencing seizure five minutes after completing the infusion of the assigned medication, the patient will be treated with an alternative second-line ASM. If the patient experiences serious treatment-related adverse effects within five minutes of the levetiracetam or phenobarbital infusion, the drug infusion will be stopped.

DETAILED DESCRIPTION:
This study will be conducted in emergency department, intensive care unit and medical wards at Yangon Children's Hospital. All children with prolonged seizures who have failed to respond to any two bolus doses of first-line benzodiazepines will be included in the study. Written informed consent will be obtained from one of the parents, guardians, or family members of children after assessing for eligibility. Parents, guardians, or family members of participants can withdrawal from the research study at any time without penalty or loss of benefits.

After selecting cases based on the inclusion criteria and obtaining written informed consent, computerized block randomization will be conducted, using a total of nine blocks to assign participants to either Group A or Group B. Group A patients will be treated with intravenous levetiracetam 40 mg/kg (maximum of 3000 mg) over 15 minutes. Group B patients will be treated with intravenous phenobarbital 20 mg/kg (maximum of 1000 mg) over 20 minutes. Injection levetiracetam will be diluted with 5% dextrose water to a concentration of 50 mg/ml. Injection phenobarbital will be diluted to become 20 ml with 5% dextrose water.

Simultaneously, detailed history and physical examination will be done according to proforma for background sociodemographic characteristics such as age, gender, seizure type and previous history of seizure. Precipitating factors to cause seizure such as fever, vomiting or diarrhoea and history suggestive of underlying aetiologies and comorbidities will also be asked. Conscious level, signs of meningism, signs of increased intracranial pressure, cardiovascular and respiratory examinations and detailed central nervous system examination will be done to find out the causes of seizure, any neurological deficits and drug side effects.

All participants will also be monitored for oxygen saturation, respiratory rate and pattern, pulse rate, pulse volume, and blood pressure to detect treatment-related adverse effects, such as acute anaphylaxis, arrhythmia, ataxia, hepatitis, hypotension, hypoxia, and respiratory depression. Monitoring will be conducted before, during, and 5 minutes after the assigned drug infusion, then hourly for 4 hours, every 2 hours for the following 4 hours, and every 4 hours thereafter.

Routine investigations such as blood for complete picture, C reactive protein, random blood sugar level and serum electrolytes or other required investigations will be tested. All participants will receive other specific treatments or supportive care, such as antibiotics and antipyretics, in accordance with ward treatment guidelines and based on any underlying diseases or comorbid conditions.

Clinical response of seizure cessation will be assessed after five minutes of injection levetiracetam or phenobarbital infusion. The primary outcome of the study will be the clinical cessation of the seizure at five minutes after the completion of the infusion of intravenous levetiracetam or phenobarbital. The secondary outcome of the study will be the recurrence of seizure within 12 hours after the commencement of the study medications, need of other medications for active seizure control within 12 hours after the commencement of the study medications, need for rapid sequence induction (RSI) with thiopentone for on-going seizure management after administration of study medications. These secondary outcomes will be assessed in treatment-responsive groups. Treatment related adverse effects will also be assessed within five minutes of drug infusion in both treatment groups and within 12 hours in treatment-responsive groups. Data analysis will be done to compare the clinical response.

If the patient's seizure has stopped five minutes after completing the infusion of the assigned medication, a maintenance dose of either levetiracetam or phenobarbital, whichever was previously used, will be administered intravenously. For group A, the maintenance dose of injection levetiracetam will be given 24 hours after the initial dose and continued twice daily, and for group B, the maintenance dose of injection phenobarbital will be given every 12 hours. It will be regarded as a response group.

If the patient is still experiencing seizure five minutes after completing the infusion of the assigned medication, the patient will be treated with an alternative second-line ASM of injection levetiracetam or phenobarbital, whichever was not previously used or diazepam infusion or midazolam infusion, following the hospital's standard protocol. It will be regarded as a failure group.

If the patient experiences serious treatment-related adverse effects within five minutes of the levetiracetam or phenobarbital infusion, the drug infusion will be stopped, and the patient will be treated with an alternative second-line ASM for seizure control, along with standard hospital protocol to manage adverse effects. It will also be regarded as a failure group due to treatment-related serious adverse effects.

After completing each block, an interim analysis will be conducted to assess efficacy and futility. To assess efficacy, Pocock's boundary method will be used, applying a consistent, adjusted p-value of approximately 0.02 (rather than the conventional 0.05) for each interim analysis to indicate early efficacy. If the conditional power falls below a pre-set threshold of 20% likelihood of achieving significance, the trial will be stopped for futility.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 1 month to 12 years with prolonged seizures who do not respond to any two bolus doses of benzodiazepines

Exclusion Criteria:

* Any of the following criteria will be excluded.

  1. Children who receive anticonvulsant treatment other than benzodiazepines for the acute management of prolonged seizures
  2. Acute symptomatic seizures due to hypertensive encephalopathy or hypoglycaemia
  3. Presence of arrythmia or respiratory depression
  4. Known case of chronic kidney disease or chronic liver disease

Ages: 1 Month to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 180 (Estimated)
Dates: Start 2025-07-22 (Actual); Primary Completion 2026-03-28 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Seizure control | at five minutes after the completion of the infusion of intravenous levetiracetam or phenobarbital
  Clinical cessation of the seizure at five minutes after the completion of the infusion of intravenous levetiracetam or phenobarbital

SECONDARY OUTCOMES:
Seizure recurrence | within 12 hours after the commencement of the study medications in treatment-responsive group
  Recurrence of seizure within 12 hours after the commencement of the study medications in treatment-responsive group
Need of other medications | within 12 hours after the commencement of the study medications in treatment-responsive group
  Need of other medications for active seizure control within 12 hours after the commencement of the study medications in treatment-responsive group
Need for rapid sequence induction (RSI) | after administration of study medications in treatment-responsive group
  Need for rapid sequence induction (RSI) with thiopentone for on-going seizure management after administration of study medications in treatment-responsive group
Treatment-related adverse effects | within five minutes of drug infusion in both treatment groups and within 12 hours in treatment-responsive groups
  Occurrence of treatment-related adverse effects within five minutes of drug infusion in both treatment groups and within 12 hours in treatment-responsive groups

CONTACTS AND LOCATIONS:
Locations (1):
- Yangon Children's Hospital, Yangon, Yangon, Burma